CLINICAL TRIAL: NCT02679599
Title: Increasing Exercise and Decreasing Sedentary Behavior Among Patients in a Cardiac Rehabilitation Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Andrew Busch, Research Scientist/Assistant Professor, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 215615
Record Dates: First submitted 2016-02-02; First posted 2016-02-10 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Acute Coronary Syndrome; Heart Failure; Other Cardiac Conditions Among Cardiac Rehabilitation Participants
MeSH Terms: conditions — Acute Coronary Syndrome; Heart Failure | interventions — Cardiac Rehabilitation

ARMS (2):
- Cardiac rehabilitation as usual (Other): Participants will receive cardiac rehabilitation as usual (i.e., as offered in the clinical setting).
  Interventions: Behavioral: Cardiac rehabilitation as usual
- Cardiac rehabilitation plus B-MOBILE-CARDIAC smartphone app (Experimental): Participants will receive cardiac rehabilitation as usual, plus access to the B-MOBILE-CARDIAC smartphone application through 4 weeks post-rehabilitation.
  Interventions: Other: B-MOBILE-CARDIAC smartphone application; Behavioral: Cardiac rehabilitation as usual

INTERVENTIONS:
Other: B-MOBILE-CARDIAC smartphone application
  Arms: Cardiac rehabilitation plus B-MOBILE-CARDIAC smartphone app
Behavioral: Cardiac rehabilitation as usual

SUMMARY:
Cardiac rehabilitation patients often fail to exercise as prescribed on days they are not attending rehabilitation and there is a steep drop off in exercise following rehabilitation completion. Moreover, little is known about the amount of time that cardiac rehabilitation patients spend in sedentary behavior, which is associated with increased risk of cardiovascular morbidity and mortality, independent of time spent in exercise. This pilot study aims to test acceptability, feasibility, and preliminary efficacy of a smartphone application (B-MOBILE-CARDIAC) for increasing time spent in moderate-to-vigorous intensity physical activity accumulated in bouts of at least 10 minutes in duration (i.e. bout-related MVPA) and decrease time spent in sedentary behavior. Up to 32 patients will be recruited, enrolled, and randomized during the first 2 weeks of cardiac rehabilitation to either: 1) B-MOBILE-CARDIAC plus cardiac rehabilitation or 2) cardiac rehabilitation alone. Participants will complete 7 days of objective activity monitoring to measure daily minutes spent in bout-related MVPA and sedentary behavior (primary outcomes) at baseline, mid-rehabilitation (6 weeks), end of cardiac rehabilitation (12 weeks), and 4-week follow-up (16 weeks). At these same time points, participants will complete questionnaires assessing sedentary behavior, MVPA, exercise tolerance, health-related quality of life, mood, and affect. At baseline and end of cardiac rehabilitation participants will undergo a blood draw to measure cardiometabolic and inflammatory risk factors and complete a test of cognitive functioning. Feasibility and acceptability of the B-MOBILE-CARDIAC application will be assessed at the 4-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. within one week of starting rehabilitation,
2. self-report that they can walk for 10 minutes without assistance from others,
3. were approved for and are planning to complete 12 weeks of rehabilitation,
4. own a compatible Android phone or are willing to be taught to use one by study staff;
5. no evidence of cognitive impairment
6. able to speak and read English,
7. aged 18-75 years,
8. no known nickel allergy, and
9. willing to follow the protocol (e.g., carry a smartphone for 16 weeks).

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-03; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change in objectively measured time engaged in sedentary behavior | Change from Baseline to 12 weeks (i.e., end of rehabilitation)
Change in objectively measured time engaged in moderate-to-vigorous intensity physical activity | Change from Baseline to 12 weeks (i.e., end of rehabilitation)

SECONDARY OUTCOMES:
Self-reported sedentary behavior (The Sedentary Behavior Questionnaire) | Baseline, 6 weeks, 12 weeks (i.e., end of rehabilitation), and 16 weeks.
Self-reported sedentary behavior (SIT-Q-7d Questionnaire) | Baseline, 6 weeks, 12 weeks (i.e., end of rehabilitation), and 16 weeks.
Self-reported physical activity (Paffenbarger Physical Activity Questionnaire) | Baseline, 6 weeks, 12 weeks (i.e., end of rehabilitation), and 16 weeks.
Self-reported exercise tolerance (Duke activity status index) | Baseline, 6 weeks, 12 weeks (i.e., end of rehabilitation), and 16 weeks.
Health related quality of life (SF-12 Health Survey) | Baseline, 6 weeks, 12 weeks (i.e., end of rehabilitation), and 16 weeks.
Depressed Mood (Patient Health Questionnaire-9) | Baseline, 6 weeks, 12 weeks (i.e., end of rehabilitation), and 16 weeks.
Affect (Positive Affect Negative Affect Scales) | Baseline, 6 weeks, 12 weeks (i.e., end of rehabilitation), and 16 weeks.
Cognitive status (Montreal Cognitive Assessment score) | Baseline and 12 weeks (i.e., end of rehabilitation).
Smartphone application acceptability (study specific scale) | Baseline through 16 weeks.
Change in objectively measured time engaged in sedentary behavior | Change from Baseline to 16 weeks
Change in objectively measured time engaged in moderate-to-vigorous intensity physical activity | Change from Baseline to 16 weeks
Lipid profile | Baseline and 12 weeks (i.e., end of rehabilitation)
C-reactive protein | Baseline and 12 weeks (i.e., end of rehabilitation)
haemoglobin A1c (HbA1C) | Baseline and 12 weeks (i.e., end of rehabilitation)
Blood pressure | Baseline, 6 weeks, 12 weeks (i.e., end of rehabilitation), and 16 weeks.
Waist circumference | Baseline, 6 weeks, 12 weeks (i.e., end of rehabilitation), and 16 weeks.
Body Mass Index (kg/m^2, weight in kilograms, height in meters) | Baseline, 6 weeks, 12 weeks (i.e., end of rehabilitation), and 16 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States